CLINICAL TRIAL: NCT06580977
Title: Exploring the Effects of Exercise on Memory and Cognition in Parkinson´s Disease
Acronym: EMCo
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Heidelberg University (Other)
Collaborators: German Foundation for Neurology (Other); University Hospital Heidelberg (Other); Universitätsmedizin Mannheim (Other); SRH Kurpfalzkrankenhaus Heidelberg (Unknown)
Responsible Party: Principal Investigator, Simon Steib, Prof. Dr., Heidelberg University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EMCo
Record Dates: First submitted 2024-05-03; First posted 2024-08-30 (Actual); Last update posted 2024-08-30 (Actual); Status verified 2024-08

CONDITIONS: Parkinson Disease
Keywords: Parkinson's Disease; rehabilitation; cardiovascular training; aerobic exercise; neuroplasticity; memory; encoding; consolidation; motor learning; acquisition; retention; cognition; sleep; brain-derived neurotrophic factor
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- cardiovascular training (Experimental): The experimental group will perform a cardiovascular training three times a week over 12 weeks.
  Interventions: Behavioral: cardiovascular training
- stretching (Active Comparator): The active control group will perform a stretching training three times a week over 12 weeks.
  Interventions: Behavioral: stretching

INTERVENTIONS:
Behavioral: cardiovascular training — Cardiovascular training will be performed in supervised sessions and in small groups of 2-5 persons at the study site. The training is performed on a cycle ergometer at 60% of peak power output (Wmax) for 30 min (i.e., 5 min warm-up, 20 min at 60% Wmax, 5 min cool-down) three times a week for twelve weeks. The exercise program will be increased by 5 min (max. 55 min) and 5% of intensity (in Watt) every two weeks. If participants report a too low (i.e., Borg scale ≤ 11) or too high (i.e., Borg scale ≥ 16) subjective rate of perceived exertion (RPE; Borg scale 6-20) intensity will be increased or decreased until the target levels are met (i.e., Borg scale 12-15). During training, heart rate, intensity (in Watt) and RPE will be monitored. Participants missing training sessions will be offered an additional week to perform up to three training sessions.
  Arms: cardiovascular training
Behavioral: stretching — The stretching training will be performed in supervised sessions and in small groups of 2-5 persons at the study site. Stretching training consists of lying, seated, and standing flexibility exercises (according to the recommendations of the American Parkinson´s Disease Foundation and the Parkinson Society Canada) for 30 min (i.e., 5 min warm-up, 20 min main part, 5 min cool-down) three times a week for twelve weeks. The exercise program will be increased by 5 min (i.e., adding additional repetitions and exercises; max. 55 min) every two weeks. Intensity of stretching exercises will be assessed by subjective rate of perceived muscle tension on a visual analog scale (VAS) from 0 to 10 and will be moderate defined as 5 to 7 on the VAS. During training VAS, heart rate, and RPE will be monitored. Participants missing training sessions will be offered an additional week to perform up to three training sessions.
  Arms: stretching

SUMMARY:
The study aims to assess the effects of cardiovascular (aerobic) training on memory formation and cognitive function in people with Parkinson's disease. Participants will be randomly allocated to one of two groups either performing cardiovascular training (experimental group) or stretching (control group) for twelve weeks, three times a week. The primary aim is to examine whether moderate-intense cardiovascular training (MICT) improves procedural memory formation (primary outcome) compared to stretching. Secondary outcomes include episodic memory formation, cognitive function, cardiorespiratory fitness, sleep quality, and brain-derived neurotrophic factor (BDNF) blood concentration levels.

DETAILED DESCRIPTION:
Besides the disabling cardinal motor symptoms, non-motor symptoms are a common clinical feature of Parkinson's disease (PD). These non-motor symptoms include, amongst others, cognitive decline and memory deficits. A growing body of evidence suggests that cardiovascular training has the potential to induce functional and structural brain changes that can translate into improved cognitive function, including memory. While data is mainly derived from studying rodents and healthy populations, cardiovascular exercise might also counteract cognitive decline and memory deficits in people with Parkinson's disease (pwPD). Therefore, the primary aim of the study is to investigate the effects of a twelve-week cardiovascular training on memory formation in pwPD.

In a randomized controlled trial, 60 persons with mild to moderate PD (i.e., Hoehn & Yahr ≤3) will either perform moderate-intensity cardiovascular training (experimental group) or stretching (control group) for twelve weeks (three times per week, totaling 36 training sessions; duration per training session 30 to 55 min). Participants will perform a procedural memory task before and after the intervention to analyze the effects on non-declarative memory formation (primary outcome). In addition, secondary and exploratory analyses will include the assessment of episodic memory formation, cognitive function, cardiorespiratory fitness, sleep quality, and BDNF blood concentration levels. The findings of the present study contribute to the current discussion on the neuroplastic effects of cardiovascular training and may have important implications for neurorehabilitation in pwPD.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed Parkinson's disease
* Disease stage ≤3 on the Hoehn & Yahr scale
* Age ranging from 50 - 80 years
* Naive to the memory tasks (primary outcomes)
* Ability to stand and walk at least 10 meters independently

Exclusion Criteria:

* Atypical Parkinsonism
* Significant level of cognitive impairment (i.e., Montreal Cognitive Assessment <21)
* Deep brain stimulation or brain pacemaker
* Diagnosed psychiatric illness
* Known clinically relevant neurological, internal or orthopedic conditions besides Parkinsonism that would interfere with the exercise paradigm
* Exceeding the recommended level of cardiovascular exercise for older adults (i.e., cardiovascular exercise done ≥150 min per week of moderate-intensity or ≥75 min per week of vigorous-intensity)

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-02-27 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Non-declarative, procedural memory (motor sequence learning) global learning score - Visuomotor Serial Targeting Task (VSTT) | Week 1-2: pre-assessment (baseline within two weeks before intervention), Week 15-16: post-assessment (within two weeks after intervention)
  To evaluate non-declarative (procedural) memory formation, a Visuomotor Serial Targeting Task (VSTT) will be used, which is widely applied to study motor sequence learning. A global motor learning score (i.e., [relative] change from start of encoding to 24h recall test) will be calculated for explicit (i.e., correct anticipatory movements defined as movements with onset times lower than in random trials and directed to the correct target [directional error at peak velocity <22°]) and implicit (i.e., spatial error to target defined as shortest distance of the movement end point from the center of the target) components of motor sequence learning and the change (delta) in the global motor learning scores from pre- to post-assessment will be analyzed. Hence, two outcome measures from the VSTT are considered to answer the primary research question: (i) change in explicit global motor learning score, and (ii) change in implicit global motor learning score from pre- to post-assessment.

SECONDARY OUTCOMES:
Non-declarative, procedural memory (motor sequence learning) encoding and consolidation - Visuomotor Serial Targeting Task (VSTT) | Week 1-2: pre-assessment (baseline within two weeks before intervention), Week 15-16: post-assessment (within two weeks after intervention)
  To evaluate the effects on the different processes of non-declarative (procedural) memory formation, the encoding (i.e., relative change in performance from beginning to end of practice) and consolidation (i.e., relative change in performance from end of practice to a 24h recall test) of the motor sequence will be investigated for the implicit and explicit components, respectively. This results in four secondary outcome variables for the VSTT: (i) change in encoding of the explicit component from pre- to post assessment; (ii) change in encoding of the implicit component from pre- to post assessment; (iii) change in consolidation of the explicit component from pre- to post assessment; (iv) change in consolidation of the implicit component from pre- to post-assessment.
Declarative, episodic memory (verbal learning) - Rey Auditory Verbal Learning Test | Week 1-2: pre-assessment (baseline within two weeks before intervention), Week 15-16: post-assessment (within two weeks after intervention)
  To evaluate the effects on declarative (episodic) memory, the German version of the Rey Auditory Verbal Learning Test will be used. Similar to non-declarative (procedural) memory (i) the change in global episodic learning score (i.e., correctly recalled words at 24 h recall test) from pre- to post-intervention will be analyzed in a first step followed by a separate analysis of (ii) the change in encoding (i.e., correctly recalled words after listening five times to the wordlist) from pre- to post-intervention and (iii) the change in consolidation (i.e., change in correctly recalled words from end of encoding to recall test) from pre- to post-intervention.
Cognitive function | Week 1-2: pre-assessment (baseline within two weeks before intervention), Week 15-16: post-assessment (within two weeks after intervention)
  To evaluate the effects on cognitive function, the domains: (i) short-term memory (Digit and Spatial Span Task forward: length of correctly reproduced sequence of digits/locations), (ii) working memory (Digit and Spatial Span Task backward: length of correctly reproduced sequence of digits/locations), (iii) inhibition (Stroop Test interference score: number of correctly named colors in the color-word condition compared to the predicted color-word score), and (vi) cognitive flexibility (Trail Making Test A & B trail flexibility score: time to complete test B compared to test A) will be assessed. A composite score including all domains to analyze change in global cognitive function from pre- to post-assessment will be calculated followed by a separate analysis of the change in the individual test scores from pre- to post-assessment.
Cardiovascular fitness | Week 1-2: pre-assessment (baseline within two weeks before intervention), Week 15-16: post-assessment (within two weeks after intervention)
  To evacuate the effects on cardiorespiratory fitness, a graded exercise test (GXT) on a cycle ergometer with spiroergometry will be performed and the change in peak oxygen consumption (VO2peak) from pre- to post intervention will be analyzed.
Objective sleep efficiency | Week 1-2: pre-assessment (baseline within two weeks before intervention), Week 15-16: post-assessment (within two weeks after intervention)
  To evaluate the effects on objective sleep quality, the change in sleep efficiency from pre- to post-assessment using wrist-worn actigraphy (ActiGraph GT9X; ActiGraph; Pensacola; USA) will be assessed.
Subjective sleep disturbance | Week 1-2: pre-assessment (baseline within two weeks before intervention), Week 15-16: post-assessment (within two weeks after intervention)
  To evaluate the effects on subjective sleep quality, the change in subjective disease-related sleep disturbance from pre- to post-assessment using the Parkinson's Disease Sleep Scale 2 (PDDS-2) total score will be assessed.
Brain-derived neurotrophic factor (BDNF) blood concentration level | Week 1-2: pre-assessment (baseline within two weeks before intervention), Week 15-16: post-assessment (within two weeks after intervention)
  To evaluate the effects on brain-derived neurotrophic factor (BDNF), serum blood samples at rest will be collected and the change from pre- to post-assessment will be analyzed.

OTHER OUTCOMES:
Non-declarative, procedural memory (motor sequence learning) further variables - Visuomotor Serial Targeting Task (VSTT) | Week 1-2: pre-assessment (baseline within two weeks before intervention), Week 15-16: post-assessment (within two weeks after intervention)
  In addition to the (a) number of correct anticipatory movements and (b) spatial error to target (i.e., primary outcomes), (i) onset time (i.e., time between target display and out movement start), (ii) movement time (i.e., time from out movement start to end), (iii) peak velocity, (iv) directional error at peak velocity (i.e., angular deviation between real and ideal movement trajectory at peak velocity), (v) spatial error to ideal movement (i.e., root mean squared error between real and ideal movement trajectory), and (vi) normalized hand-path area (i.e., area enclosed by the out and in movement divided by the squared path length) will be inspected to analyze practice-related changes in temporal and kinematic movement characteristics.
Sociodemographic & physical characteristics | Week 1-2: pre-assessment (baseline within two weeks before intervention), Week 15-16: post-assessment (within two weeks after intervention)
  1. Age, biological sex
  2. Years of education
  3. Height, weight, body mass index
  4. Handedness (Edinburgh Handedness Inventory)
Non-motor symptoms (nonmotor experiences of daily living) - Movement Disorder Society Unified Parkinson's Disease Rating Scale Part I | Week 1-2: pre-assessment (baseline within two weeks before intervention), Week 15-16: post-assessment (within two weeks after intervention)
  Movement Disorder Society Unified Parkinson's Disease Rating Scale (UPDRS) Part I total score (0-52)
Motor symptoms (motor examination) - Movement Disorder Society Unified Parkinson's Disease Rating Scale Part III | Week 1-2: pre-assessment (baseline within two weeks before intervention), Week 15-16: post-assessment (within two weeks after intervention)
  Movement Disorder Society Unified Parkinson's Disease Rating Scale (UPDRS) Part III total score (0-132)
Total daily medication - Levodopa equivalent daily dose | Week 1-2: pre-assessment (baseline within two weeks before intervention), Week 15-16: post-assessment (within two weeks after intervention)
  Total levodopa equivalent daily dose (LEDD) in mg
Cognitive status - Montreal Cognitive Assessment | Week 1-2: pre-assessment (baseline within two weeks before intervention), Week 15-16: post-assessment (within two weeks after intervention)
  Montreal Cognitive Assessment (MoCA) total score (0-30 points)
Quality of life - Parkinson´s Disease Questionnaire-39 | Week 1-2: pre-assessment (baseline within two weeks before intervention), Week 15-16: post-assessment (within two weeks after intervention)
  Parkinson´s Disease Questionnaire-39 (PDQ-39) dimension scores (0-100) and total score (0-100)
Objective sleep quality | Week 1-2: pre-assessment (baseline within two weeks before intervention), Week 15-16: post-assessment (within two weeks after intervention)
  Actigraphy (wrist-worn accelerometer for seven days and nights): sleep onset latency, total sleep time, wake after sleep onset, number of awakenings
Subjective sleep quality | Week 1-2: pre-assessment (baseline within two weeks before intervention), Week 15-16: post-assessment (within two weeks after intervention)
  Pittsburgh Sleep Quality Index (PSQI) total score (0-21 points)
Daytime sleepiness | Week 1-2: pre-assessment (baseline within two weeks before intervention), Week 15-16: post-assessment (within two weeks after intervention)
  Epworth Sleepiness Scale (ESS) total score (0-10 points)
Severity of depression - Beck Depression Inventory | Week 1-2: pre-assessment (baseline within two weeks before intervention), Week 15-16: post-assessment (within two weeks after intervention)
  Beck Depression Inventory (BDI) total score (0-63)
Severity of anxiety - Beck Anxiety Index | Week 1-2: pre-assessment (baseline within two weeks before intervention), Week 15-16: post-assessment (within two weeks after intervention)
  Beck Anxiety Index (BAI) total score (0-63)
Objective physical activity | Week 1-2: pre-assessment (baseline within two weeks before intervention), Week 15-16: post-assessment (within two weeks after intervention)
  Actigraphy (wrist-worn accelerometer for seven days): total volume of physical activity, steps per day, minutes spent at different intensity levels, total daily vector magnitude counts
Subjective physical activity last week | Week 1-2: pre-assessment (baseline within two weeks before intervention), Week 15-16: post-assessment (within two weeks after intervention)
  International Physical Activity Questionnaire (IPAQ) - short form: MET hours per week
Subjective physical activity last four weeks | Week 1-2: pre-assessment (baseline within two weeks before intervention), Week 15-16: post-assessment (within two weeks after intervention)
  German Physical Activity Questionnaire 50+ (German PAQ 50+): MET hours per week

CONTACTS AND LOCATIONS:
Overall Officials: Simon Steib, Prof. Dr., Principal Investigator — Heidelberg University; Philipp Wanner, Dr., Principal Investigator — Heidelberg University
Locations (1):
- Heidelberg University, Heidelberg, Baden-Wurttemberg, Germany

IPD SHARING:
Plan to Share IPD: Yes
The anonymized data will be shared after completion of the study and publication of the primary results (presumably via OpenScienceFramework - OSF; https://osf.io/).
Supporting Information: Study Protocol, SAP
Time Frame: After completion of the study and publication of the primary outcome for at least ten years
Access Criteria: open data (presumably CC-BY Attribution 4.0 International licence)

REFERENCES:
- See also: Project website — https://www.issw.uni-heidelberg.de/arbeitsbereiche/but/projekte.html

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-04-21): https://cdn.clinicaltrials.gov/large-docs/77/NCT06580977/Prot_SAP_000.pdf